CLINICAL TRIAL: NCT00120731
Title: Urinary Chemistry and Acid-Base Effects of Potassium Citrate in Children With Idiopathic Hypercalciuria and Urolithiasis
Brief Title: Effects of Potassium Citrate in Urine of Children With Elevated Calcium in Urine and Kidney Stones
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Determined not feasible
Sponsor: Children's Mercy Hospital Kansas City (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG#05036
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Kidney Calculi
Keywords: Recurrent nephrolithiasis; Potassium Citrate; Hypercalciuria; Distal Renal Tubular Acidosis; Nephrolithiasis in children
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Hypercalciuria; Acidosis, Renal Tubular | interventions — Potassium Citrate; Acetazolamide; Oxalates; Purines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Potassium Citrate
Drug: Acetazolamide
Behavioral: Diet low in oxalate and purines

SUMMARY:
High amounts of calcium in the urine (hypercalciuria) can cause development of kidney stones in children. Treatment for these children includes plenty of fluids, a low-salt diet and medications such as potassium citrate. A major advantage of potassium citrate, as compared to hydrochlorothiazide, is its lack of side effects. One problem the researchers and others have observed is that some children continue to form kidney stones despite correction of hypercalciuria with potassium citrate. One possible explanation is that in some individuals potassium citrate therapy results in an excessive elevation of urine pH, a situation that may predispose to calcium phosphate stone formation. In this study, the researchers will study the effects of potassium citrate on urine chemistries and acid-base balance in three groups of children aged 5-17 years:

* children who are hypercalciuric stone formers;
* healthy children without a history of hypercalciuria or kidney stones.

Particular attention will be paid to try to identify those who develop a very high urine pH (>8) and the factors leading to this metabolic reaction.

The researchers will try to learn whether it is the child's characteristics, the disease manifestations, the dose of the drug, or a combination of the above which may be the cause of the development of very alkaline urine. Based on the results, the researchers hope to be able to better "tailor" the individual treatment for each child with kidney stones.

DETAILED DESCRIPTION:
Hypercalciuria is a common clinical pediatric problem that in some children is associated with renal stones. Most renal stones (80%) are formed by calcium oxalate, calcium phosphate phases (apatite), and brushite (calcium monohydrogen phosphate). Hypercalciuria can be either primary (accounts for the vast majority of children with calcium stones) or secondary. Treatment for children with calcium stones involves non-pharmacological and pharmacological interventions. Non-pharmacological interventions include high fluid intake, low sodium, and potassium enhanced diet, with RDA calcium and protein. Historically, the specific treatment for hypercalciuric stone formers has included thiazides, which reduce calciuria, lower the urinary saturation of calcium oxalate and phosphate, and restore normal intestinal calcium absorption. However thiazides induce hypokalemia and hypocitraturia, and the latter attenuates the beneficial effects of the drug on stone formation. Currently, the drug of choice replacing thiazides in treating idiopathic hypercalciuria is potassium citrate. Potassium citrate is readily absorbed from the gastrointestinal tract, and after being excreted in the urine, it inhibits the crystallization of stone forming calcium salts by binding the calcium ion, thus decreasing its urinary saturation and inhibiting the nucleation and crystal growth of calcium oxalate; therefore, potassium citrate is an effective stone inhibitor agent. A major advantage of potassium citrate is its lack of side effects. One of the problems seen in clinical practice is that some children with primary hypercalciuria, even after the calciuria is treated successfully with potassium citrate, continue to develop stones. It has been suggested that an elevation in urine pH, seen in some patients treated with potassium citrate, may result in an alkaline urinary milieu which promotes calcium phosphate stone formation. In this study, the researchers plan to investigate the effects of potassium citrate on urine chemistries and acid-base balance in children who are hypercalciuric stone formers. The researchers will try to identify whether the beneficial effects of potassium citrate supplementation on lowering urine calcium and increasing citrate might be offset by too high urine pH (>8) which could promote the formation of calcium phosphate stones. Three groups of subjects aged 5-17 years will be studied: group 1 - idiopathic hypercalciuric stone formers; group 2 - idiopathic hypercalciuric non-stone formers; and group 3 - normocalciuric subjects. Three visits will be scheduled for each participant, and the subjects will receive two doses of potassium citrate. Urine chemistries and acid-base parameters will be measured. The researchers will try to learn whether it is the child's characteristics, the disease manifestations, the dose of the drug, or a combination of the above which may be the cause of the development of very alkaline urine. Based on the study results, the researchers hope to be able to better "tailor" the individual treatment for each child with kidney stones due to idiopathic hypercalciuria.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-17 years with idiopathic hypercalciuria who have history of kidney stones.
* Healthy children aged 5-17 years without a history of hypercalciuria or kidney stones.

Exclusion Criteria:

* Children with urolithiasis secondary to metabolic disorders unrelated to hypercalciuria (e.g. oxaluria, hypocitraturia, cystinuria), or due to secondary causes of calciuria (hypercalcemia, hyperparathyroidism, corticosteroids, furosemide).
* Children with renal insufficiency, active urinary tract infection, hyperkalemia, gastrointestinal diseases, heart failure.
* Children who receive angiotensin-converting enzyme inhibitors, anticholinergic medications or digitalis.
* Children who cannot safely stop receiving the prohibited concomitant medications due to other underlying medical conditions

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Changes in urine pH, citrate, calcium and bicarbonate after treatment with increasing doses of potassium citrate | Duration of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ari Auron, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Tapaneya-Olarn W, Khositseth S, Tapaneya-Olarn C, Teerakarnjana N, Chaichanajarernkul U, Stitchantrakul W, Petchthong T. The optimal dose of potassium citrate in the treatment of children with distal renal tubular acidosis. J Med Assoc Thai. 2002 Nov;85 Suppl 4:S1143-9. PMID 12549788